CLINICAL TRIAL: NCT00710307
Title: Descriptive, Cross-sectional and Prospective Epidemiology Study, on the Identification of Insulin-like Growth Factor-1 Status in Idiopathic Short Stature Children (EPIGROW Study)
Brief Title: Epidemiology Study on Insulin-like Growth Factor-1 in Children With Idiopathic Short Stature (EPIGROW Study)
Acronym: EPIGROW
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 2-79-52800-001
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Idiopathic Short Stature
MeSH Terms: interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood will be collected. The blood sample will be kept as long as necessary and for a maximum of 5 years.

INTERVENTIONS:
Procedure: Blood sampling — Blood samples will be collected at visit 1 (day 1) and at visit 2 (day 14 to 45).
Genetic: Genetic analysis — The sample for genetic analyses may be taken at Visit 1. The blood sample volume will be 6 mL.

SUMMARY:
The purpose of the protocol is to describe the distribution of IGF-1 deficiency in the studied population of Idiopathic Short Children without Growth Hormone Deficiency or any other identified cause of short stature and not treated with recombinant Growth Hormone or IGF-1

ELIGIBILITY:
Inclusion Criteria:

* Short children, height ≤ -2.5 SDS
* Age ≥ 2 years
* With at least one normal or elevated peak GH response to a stimulatory test (peak GH ≥ 7 ng/mL) at the time of the study and/or at a given time-point during the last 12 months
* Pre-pubertal
* Signed Informed Consent, including agreement to have blood samples taken for hormonal measurement and genetic analysis, by both parents or by Legally Acceptable Representatives when applicable and the child when applicable

Exclusion Criteria:

* The following identified causes of short stature:
* GH-deficient short stature
* Other endocrine causes (hypothyroidism, Cushing's syndrome, parathyroid or vitamin D disorders, hypogonadism)
* Identified syndromes with genetic abnormalities (including Turner, Noonan and Russell-Silver syndromes)
* Chronic diseases including malnutrition, coeliac disease, chronic inflammation, muscular dystrophy, thalassaemia, blood disorders, severe liver or kidney disease and severe cyanotic heart disease
* Chronic diseases requiring treatment with chronically administered corticosteroids
* Skeletal dysplasia
* Psychosocial short stature
* Patients having received irradiation, including total body irradiation
* Patients currently on GH or IGF-1 therapy or having received GH or IGF-1 therapy in the last 12 months
* Patients likely to require GH, IGF-1 or chronic corticosteroid treatment during the study
* Any mental condition that prevents both parents or Legally Acceptable Representatives and the child when applicable from understanding the nature, scope and possible consequences of the study, or any evidence of an uncooperative attitude

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Idiopathic Short Stature children
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a mean of the two basal IGF-1 measurements ≤-2.0 SDS, > -2.0 SDS and below 0 SDS, ≥ 0.0 SDS | Day 1 for the first sample; between Day 14 and Day 45 for the second sample

SECONDARY OUTCOMES:
Proportion of patients with height ≤ -3.0 SDS,and height > -3.0 SDS and ≤ -2.5 SDS | Day 1
Description of mean basal IGF-1 and IGFBP-3 levels, and basal ALS and prolactin levels in patients with height ≤ -3.0 SDS, and height > -3.0 SDS and ≤ -2.5 SDS | Day 1 and Day 14-45
Proportion of patients having presented at least one historical documented clinically significant episode of hypoglycaemia | Before the start of the study and during the study.
Identification of candidate genes and/or DNA aberrations or changes potentially associated with short stature. DNA regions identified during the genome-wide scan will be further mapped at higher resolution (DNA-sequencing) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Paris, France